CLINICAL TRIAL: NCT03716141
Title: Autologous Platelets Rich Plasma (APRP) Treatment Vs Saline Dressing for the Management of Diabetic Foot Ulcer
Acronym: APRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, principal investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s6
Record Dates: First submitted 2018-07-11; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Platelets Rich Plasma (Active Comparator): In this group we will be managing diabetic wounds with platelet rich plasma treatment.
  Interventions: Other: Autologous Platelets Rich Plasma Treatment
- Conventional Saline dressing (Active Comparator): In this group we will be managing diabetic wounds with normal saline dressing.
  Interventions: Other: Conventional Saline dressing

INTERVENTIONS:
Other: Autologous Platelets Rich Plasma Treatment — For PRP preparation 10 mL of the patient blood was collected. The blood was centrifuged at 2000 rpm for 5 min to obtain plasma. Then, this plasma was centrifuged at 3000 rpm for another 5 min to collect platelets. Platelets were diluted in 5 mL plasma to form PRP.
  Arms: Autologous Platelets Rich Plasma
Other: Conventional Saline dressing — saline dressing of diabetic wounds will be done
  Arms: Conventional Saline dressing

SUMMARY:
The aim of this study is to compare between the platelet rich plasma and normal saline dressing in the healing diabetic foot ulcers. It will be a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot wound less than 5cm in greatest diameter Non healing duration greater than 3 months Non infected Palpable distal pulses

Exclusion Criteria:

* Infected wound Wound greater than 5 cm Patient having HBa1c greater than 8% Renal failure Wound with bone exposed or having osteomyelitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 8 to 12 weeks
  complete healing of diabetic foot

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided